CLINICAL TRIAL: NCT03287297
Title: Association Between Dietary Habits and Gestational Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mokhtar Abdel-Hameed, Principal investigator, Assiut University
Other Study IDs: 17100275
Record Dates: First submitted 2017-09-16; First posted 2017-09-19 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OGTT & HBA1c — oral glucose tolerance test & HBA1c: by measuring glycated hemoglobin

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as carbohydrate intolerance of varying severity with onset or first recognition during pregnancy. The diagnosis of gestational diabetes is important, because of the increased risk of adverse maternal and feto-neonatal outcomes. In addition, GDM also confers a future risk of type 2 diabetes to mothers and their fetus. Dietary components associated with GDM risk include macronutrients, micronutrients, and individual foods, such as refined carbohydrates, saturated fats, soft drinks and processed meats. The Pre-pregnancy dietary patterns may affect women risk of developing GDM. A diet high in red and processed meat was associated with a significantly elevated risk.

DETAILED DESCRIPTION:
*Aim of the work: To investigate associations between maternal dietary patterns and GDM.

* Patients and Methods:

  * Study design: A cross sectional study was conducted.
  * Study site: GDM Outpatient Clinic of Assiut University Hospital.
  * Study population: The study will include all pregnant women at 24th to 28th gestational age, who attending to GDM Outpatient Clinic during the period of The Study.
  * Inclusion criteria include pregnant women at 24th to 28th age of gestation.
  * Exclusion criteria include pre-gestational diabetic women and pregnant women before and after 24th -28th week of gestation.
  * Instrument: Structured designed questionnaire: Which consists of socio-demographic characteristics, Medical and obstetric history and other risk factors for GDM including previous GDM, family history of diabetes, twins in current pregnancy, history of PCO and macrosomic baby in current or previous pregnancy, also contains information about regularity and frequencies of daily meals taken by the women, and information about food group frequencies per week, food groups like vegetables, fruits, fast food , red and processed meat, fish and seafood, whole grains, cereal fiber, sweetened beverage, dessert food and use of multivitamins.
  * Data collection: Direct interview will be done with each participant separately for filling the food frequency questionnaire by the researcher himself during the period from January 2017 to June 2017
* Clinical examination:

  * BP (mmHg)
  * Pulse
  * Body Weight (kg)
  * Height (cm)
  * BMI

Laboratory Examination

* OGTT (75gm) 2hr
* HBA1c (if Bl. Glucose ≥ 200mg/dl).

ELIGIBILITY:
Inclusion Criteria:

* include pregnant women at 24th to 28th age of gestation.

Exclusion Criteria:

* include pre-gestational diabetic women and pregnant women before and after 24th -28th week of gestation.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study will include all pregnant women at 24th to 28th gestational age
Study Population: The study will include all pregnant women at 24th to 28th gestational age, who attending to GDM Outpatient Clinic.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Level | Baseline
  Mean difference In Blood Glucose Level Among Cases

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alfadhli EM. Gestational diabetes mellitus. Saudi Med J. 2015 Apr;36(4):399-406. doi: 10.15537/smj.2015.4.10307. PMID 25828275
- [Background] Bhatt AA, Dhore PB, Purandare VB, Sayyad MG, Mandal MK, Unnikrishnan AG. Gestational diabetes mellitus in rural population of Western India - Results of a community survey. Indian J Endocrinol Metab. 2015 Jul-Aug;19(4):507-10. doi: 10.4103/2230-8210.159061. PMID 26180767
- [Background] Kampmann U, Madsen LR, Skajaa GO, Iversen DS, Moeller N, Ovesen P. Gestational diabetes: A clinical update. World J Diabetes. 2015 Jul 25;6(8):1065-72. doi: 10.4239/wjd.v6.i8.1065. PMID 26240703
- [Background] Poomalar GK, Rangaswamy V. A comparison of fasting plasma glucose and glucose challenge test for screening of gestational diabetes mellitus. J Obstet Gynaecol. 2013 Jul;33(5):447-50. doi: 10.3109/01443615.2013.771156. PMID 23815193
- [Background] Agarwal MM. Gestational diabetes mellitus: An update on the current international diagnostic criteria. World J Diabetes. 2015 Jun 25;6(6):782-91. doi: 10.4239/wjd.v6.i6.782. PMID 26131321
- [Background] Ovesen PG, Jensen DM, Damm P, Rasmussen S, Kesmodel US. Maternal and neonatal outcomes in pregnancies complicated by gestational diabetes. a nation-wide study. J Matern Fetal Neonatal Med. 2015;28(14):1720-4. doi: 10.3109/14767058.2014.966677. Epub 2015 Jan 8. PMID 25228278
- [Background] Seshiah V; Diabetes in Pregnancy Study Group. Fifth National Conference of Diabetes in Pregnancy Study Group, India. J Assoc Physicians India. 2010 May;58:329-30. No abstract available. PMID 21117358
- [Background] Zhang C, Ning Y. Effect of dietary and lifestyle factors on the risk of gestational diabetes: review of epidemiologic evidence. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1975S-1979S. doi: 10.3945/ajcn.110.001032. Epub 2011 May 25. PMID 21613563
- [Background] Zhang C, Schulze MB, Solomon CG, Hu FB. A prospective study of dietary patterns, meat intake and the risk of gestational diabetes mellitus. Diabetologia. 2006 Nov;49(11):2604-13. doi: 10.1007/s00125-006-0422-1. Epub 2006 Sep 7. PMID 16957814
- [Background] Qiu C, Zhang C, Gelaye B, Enquobahrie DA, Frederick IO, Williams MA. Gestational diabetes mellitus in relation to maternal dietary heme iron and nonheme iron intake. Diabetes Care. 2011 Jul;34(7):1564-9. doi: 10.2337/dc11-0135. PMID 21709295